CLINICAL TRIAL: NCT05134818
Title: Use of an Observer Tool to Improve Learning Outcomes of Incoming Anesthesia Residents During Procedural Simulation Training of Central Venous Catheter Insertion: a Randomized Controlled Trial of Simulation Training
Brief Title: Observer Tool Use and Learning Outcomes for Central Venous Catheter Insertion Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université Paris-Sud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LabForSims-004
Record Dates: First submitted 2021-10-29; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Education; Simulation
Keywords: simulation; education; observer tool; central venous catheter

STUDY DESIGN:
Intervention Model Description: Parallel assignment, not blinded, randomized study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group OT + (Experimental): In this group (OT +), the resident will complete an observer tool each time another resident is observed to insert a CVC on the simulator.
  Interventions: Other: observer tool
- group OT- (No Intervention): In this group (OT-), the resident will not use the observer tool and will observe other residents to insert a CVC on the simulator without any physical support.

INTERVENTIONS:
Other: observer tool — comparison of the efficacy of an observer tool to enhance learning of technical skills of CVC insertion in anesthesiology residents The resident will complete an observer tool each time another resident is observed to insert a CVC on the simulator.
  Arms: group OT +

SUMMARY:
Learning to insert a central venous catheter (CVC) is essential in anesthesiology and the use of simulation is recommended. Since 2017, this training has been integrated into the curriculum for incoming first year anesthesia residents in Île de France and combines a theoretical part (flipped classroom) and a practical part on a simulator. Given the large number of residents, the time to teach the procedure during the simulation session is limited. To increase the positive effects of the simulation when the learner is in the role of observer, some authors have proposed to strengthen the educational effect through the use of an observer tool that observers must complete by analyzing the progress of the task performed by their colleagues. This is a list describing the set of key points to be achieved. However, data concerning the educational value of these observer tools are limited. Studies on the use of these tools during crisis management training in the operating room assessed by high-fidelity simulation has been already conducted but not on their use during procedural simulation.

The objective of this study will be to assess the value of using an observer tool (OT) (including the key points during the insertion of an internal jugular CVC) to improve learning outcomes of incoming anesthesia residents during procedural simulation training.

DETAILED DESCRIPTION:
Learning to insert a central venous catheter (CVC) is essential in anesthesiology and the use of simulation is recommended. Since 2017, this training has been integrated into the curriculum for incoming first year anesthesia residents in Île de France and combines a theoretical part (flipped classroom) and a practical part on a simulator. Given the large number of residents, the time to teach the procedure during the simulation session is limited. To increase the positive effects of the simulation when the learner is in the role of observer, some authors have proposed to strengthen the educational effect through the use of an observer tool that observers must complete by analyzing the progress of the task performed by their colleagues (2). This is a list describing the set of key points to be achieved. However, data concerning the educational value of these observer tools are limited. Studies on the use of these tools during crisis management training in the operating room assessed by high-fidelity simulation has been already conducted but not on their use during procedural simulation.

The objective of this study will be to assess the value of using an observer tool (OT) (including the key points during the insertion of an internal jugular CVC) to improve learning outcomes of incoming anesthesia residents during procedural simulation training.

This prospective and randomized study will be performed in the simulation center of Paris-Saclay University (LabForSIMS). This training takes place annually at the beginning of the first six-month rotation during an initial training seminar ("bootcamp"). All incoming residents (approximately 90 residents / year) participate on a mandatory basis.

Each CVC insertion training session includes a theoretical part carried out in the form of flipped classroom (sending pedagogical documents upstream) and a practical part on a simulator. Each practical session (1h30, about 7 residents/1 instructor) is repeated twice during the half-day. The workshop has three stages: theoretical reminder, supervised practice on echogenic gelatin to learn needling under ultrasound, then supervised practice on a CVC simulator (part task chest trainer allowing ultrasound visualization) for the insertion of CVC. Each resident trains at least once on this simulator and is an observer of the other training sessions.

After informed consent, residents will be included. Each session will be randomized upstream by:

* Group with observer tool (OT +) during practical training on a simulator
* Group without observer tool (OT-) The observer tool used will be adapted from a previously published checklist which includes the main items to be carried out when inserting a CVC. It will be completed by residents from the OT + group each time another resident is observed. It will only be used to reinforce learning and will not be used for summative evaluation.

The primary outcome will be a composite score describing acquisition of the CVC procedural skills immediately after training by comparing the groups using or not the OT (level 1-2-3 of the Kirkpatrick model). The composite score (used in one of our previous studies [Blanié A et al. 2021 submitted]) includes: knowledge MCQs (/ 20), perception of practical (/ 10) and theoretical (/ 10) improvement of knowledge and skills, perception of the future professional impact of this training (/ 10) and satisfaction with the training session (/ 10). All items scored out of 10 will be measured by a Likert scale from 0 to 10.

The secondary outcomes will include separate analysis of each item of the composite score. Moreover, initial retention will be analyzed at 1 month, using the same items as above. Evaluation of professional practice will also be recorded by the resident during the 1st month after the training and will include the number of CVCs placed and for each CVC insertion via the internal jugular route (for the first 5): the number of punctures, success or failure, complications (pneumothorax, arterial puncture, others) (level 3 and 4 of the Kirkpatrick model).

A reminder will be sent every two weeks and a medical book will be offered to each resident who will have fully completed the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* first year anesthesiology residents

Exclusion Criteria:

* absence to the CVC training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
composite score describing acquisition of the CVC procedural skills using a questionnaire immediately after training | 10 minutes at the end of the session
  The questionnaire of the composite score includes : 20 knowledge MCQs (/ 20), questions about the perception of practical (0 to 10) and theoretical (0 to 10) improvement of knowledge and skills, perception of the future professional impact of this training (0 to 10) and satisfaction with the training session (0 to 10). All items scored out of 10 will be measured by a Likert scale from 0 to 10.

SECONDARY OUTCOMES:
question of each item of the composite score | 10 minutes at the end of the session
  Separate analysis of each question of the composite score: knowledge MCQs (/ 20), perception of practical (0 to 10) and theoretical (0 to 10) improvement of knowledge and skills, perception of the future professional impact of this training (0 to 10) and satisfaction with the training session (0 to 10).
retention using a questionnaire by e-mail (self-report) | 10 minutes at 1 month
  initial retention analyzed at 1 month, using the same questionnaire as above (the composite score includes : 20 knowledge MCQs (/ 20), questions about the perception of practical (0 to 10) and theoretical (0 to 10) improvement of knowledge and skills, perception of the future professional impact of this training (0 to 10) and satisfaction with the training session (0 to 10). All items scored out of 10 will be measured by a Likert scale from 0 to 10)
Evaluation of professional practice using a questionnaire by e-mail (self-report) | 1 minutes during the first month after
  Evaluation of professional practice will also be recorded by the resident during the 1st month after the training using a questionnaire send by e-mail (self-report) (level 3 and 4 of the Kirkpatrick model). It will include a question of the number of CVCs placed (0 to >10).
Evaluation of professional practice using a questionnaire by e-mail (self-report) | 2 minutes during the first month after
  Evaluation of professional practice will also be recorded by the resident during the 1st month after the training using a questionnaire send by e-mail (self-report) (level 3 and 4 of the Kirkpatrick model). It will include questions for each CVC insertion via the internal jugular route (for the first 5) about the number of punctures (0 to >10), success or failure, complications (pneumothorax, arterial puncture, others) (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Blanié, MD, PhD, Principal Investigator — SRP07 UNIVERSITE PARIS-SACLAY
Locations (1):
- Faculté de médecine Paris Sud, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No